CLINICAL TRIAL: NCT01873599
Title: Impact of an Online Positive Affect Journaling Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Penn State University (Other)
Responsible Party: Principal Investigator, Christopher Sciamanna, MD, MPH, Chief, Division of General Internal Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 41160EP
Record Dates: First submitted 2013-06-05; First posted 2013-06-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention condition will be asked to write for 15 minutes on three days each week to one of the seven positive affect writing prompts on www.stressvax.com. Subjects who do not complete a journal entry within 7 days will receive an email reminder, in case they have lost their password or have some technical problem accessing the site.
  Interventions: Behavioral: Positive Affect Journaling
- Control (No Intervention): As there is no clinical standard of care treatment for psychological distress, patients randomized into this condition will receive their usual care. At the end of three months, subjects in this condition will be given access to the positive affect journaling intervention.

INTERVENTIONS:
Behavioral: Positive Affect Journaling
  Arms: Intervention

SUMMARY:
In this study the investigators plan to recruit 70 patients reporting high levels of stress to test the impact of Positive Affect Journaling. Patients randomized to use the online intervention will be asked to journal about one of seven topics, several days each week, for three months. The topics (e.g., "What went well") are designed to help the individual focus on some positive aspect of their life or themselves over the past day. Each topic is based on prompts shown to be effective in studies of up to one week in duration. In the summer of 2012, our research team pilot tested each prompt with 20 patients with high levels of anxiety, which led to important changes to the prompts, to increase their potential impact. The main aim is to understand the impact of Positive Affect Journaling on psychological distress, as measured by the National Health Interview Survey.

ELIGIBILITY:
Inclusion Criteria:

* Fluently speaks, writes, and read English
* Report elevated levels of stress
* Be between 21-80 years of age
* Have access to the Internet
* Have an ECOG Performance Status of 0 (Fully active) through 3 (Limited self-care)

Exclusion Criteria:

* High risk for suicidality on the Structured Clinical Interview for DSM Disorders (SCID).
* Pregnant or planning to get pregnant in the next 3 months
* Moving in the next 6 months

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
National Health Interview Survey | 3 month follow up
  The NHIS measures perceived levels of stress over the past 12 months.

SECONDARY OUTCOMES:
Brief Resilience Scale | 3 month follow up
  The BRS is a 6-item self-report measure of perceived resilience, including items such as "It does not take me long to recover from a stressful event" The BRS has high levels of internal consistency, with Cronbach's alpha ranging from .80-.91
Perceived Stress Scale | 3 month follow up
  The PSS consists of 10 items that assess perceived stress. The items are scored on a 4-point scale (45). The measure demonstrates strong internal consistency with a Cronbach's alpha of .88
Satisfaction with Life scale | 3 month follow up
  The SWL is a five-item scale that assesses overall life satisfaction. The SWL has a 2-month test-retest reliability of 0.82 and a Cronbach's alpha of 0.87
Social Provisions Scale | 3 month follow up
  The SPS assesses the extent to which one perceives their social relationships to be supportive. This 24-item measure has a Cronbach's alpha of 0.91
Healthy Days score | 3 month follow up
  Created by the Centers for Disease Control, this measure assesses the number of days of poor mental health, physical health, poor sleep and other symptoms, as well as overall health
Positive and Negative Affect Schedule score | 3 month follow up
  The 20-item PANAS consists of two subscales, in which respondents indicate the extent to which they felt specific positive and negative emotions over a specific time frame. Internal consistencies are high (Crohnbach's alpha = 0.85-0.88)
Cancer Quality of Life | 3 month follow up
  The EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sciamanna, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Smyth JM, Johnson JA, Auer BJ, Lehman E, Talamo G, Sciamanna CN. Online Positive Affect Journaling in the Improvement of Mental Distress and Well-Being in General Medical Patients With Elevated Anxiety Symptoms: A Preliminary Randomized Controlled Trial. JMIR Ment Health. 2018 Dec 10;5(4):e11290. doi: 10.2196/11290. PMID 30530460